CLINICAL TRIAL: NCT02837185
Title: Physiological Effects of Botulinum Toxin Therapy in Primary Cervical Dystonia
Brief Title: Effects of Botulinum Toxin on Muscle and Brain Activity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit controls and limited research staff to complete project.
Sponsor: University of Florida (Other)
Collaborators: Dystonia Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201600759
Record Dates: First submitted 2016-07-07; First posted 2016-07-19 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Cervical Dystonia, Primary
Keywords: Cervical dystonia; Transcranial magnetic stimulation; Electromyography; TMS; EMG
MeSH Terms: conditions — Cervical Dystonia, Primary; Torticollis | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cervical Dystonia (Experimental): 'Botulinum Toxin injection' will be done and 'physiological measures' will then be collected.
  Interventions: Procedure: Botulinum Toxin injection; Other: Physiological measures
- Healthy controls (Other): No Botulinum toxin is injected, 'physiological measures' will be collected as a healthy comparator.
  Interventions: Other: Physiological measures

INTERVENTIONS:
Procedure: Botulinum Toxin injection — Botulinum toxin injection for cervical dystonia subjects (as part of clinical care)
  Arms: Cervical Dystonia
Other: Physiological measures — These include TMS and EMG measurements

SUMMARY:
This study will look into the effects of Botulinum Toxin in patients with primary cervical dystonia. The effects will be determined by neck muscle activity measurements and brain function activity measurements. The goal of the study is to try to identify markers of the effects of Botulinum toxin.

DETAILED DESCRIPTION:
Primary Cervical Dystonia (PCD) is the most common type of focal dystonia. In addition to pain, PCD is associated with disability in many activities of daily living; social stigma and embarrassment; and decreased quality of life. Botulinum toxin (BoNT) therapy is the "gold standard" for treatment of PCD. Although effective in improving dystonia symptoms, BoNT injections have been associated with suboptimal improvements and the benefits of BoNT may last shorter than the expected time frame of 12 weeks. PCD subjects are referred for deep brain stimulation surgery if there is poor or inconsistent response to medical treatment. In addition to the need for repetitive injections, subjects may suffer from side effects such as neck pain, muscle weakness, head drop, breathing difficulty, and swallowing issues. BoNT therapy outcomes are not likely to improve until and unless the investigators understand the underlying mechanisms of action.

The primary goal of this study is to examine the physiological effects of BoNT therapy and to advance the understanding of the pathophysiology of dystonia. BoNT therapy is commonly perceived to induce peripheral muscle weakness through inhibition of acetylcholine release at the neuromuscular junction. However many argue that this is not likely the only or primary mechanism of action, as many subjects have improvement in dystonia without discernible muscle weakness and others have significant weakness and no improvement in their dystonia. Indeed, BoNT has been proposed to induce central effects possibly related to modulation of the muscle spindle afferent feedback or a retrograde transport of toxin to the central nervous system. A leading theory underpinning the pathophysiology of dystonia is loss of motor inhibition (or increased excitability) at the level of the spinal cord, brainstem and the motor cortex. Thus, modulation of pathology in these central pathways is critical for control of dystonia. Transcranial magnetic stimulation (TMS) is a noninvasive physiological technique for assessment of motor cortex excitability. Paired-pulse TMS paradigms, such as short-interval intracortical inhibition (SICI) and intracortical facilitation (ICF) are well established paradigms for evaluation of motor cortex excitability.

SICI is measured by delivering a subthreshold conditioning pulse prior to the suprathreshold test pulse at short interstimulus intervals (ISI) of 1-5 milliseconds (ms) resulting in a lower motor evoked potential (MEP) response to the test pulse. SICI is regarded as a gamma-aminobutyric acid A (GABA-A) receptor-mediated inhibition that involves activation of the cortical inhibitory interneurons. ICF is measured using a paradigm similar to SICI but with a longer ISI of 8-30 ms resulting in increase in MEP response. Glutamate is probably involved in producing ICF through cortical facilitation.

In focal dystonia, including PCD, there is failure of SICI recorded from hand muscles, and conversely, there is enhanced ICF recorded from hand muscles. These paradigms were not recorded from neck muscles as they are technically challenging. Nevertheless an important finding was noted that in PCD, the motor cortical inhibition is widespread and extends beyond the area of symptomatic muscles.

TMS was used to assess the effects of BoNT on SICI in subjects with arm dystonia. SICI in distal hand muscle increases at one month after BoNT injections and returns to the previously abnormal levels of excitability at three months. It can be speculated that the BoNT therapy to arm muscles modulates the afferent input from muscles, which probably results in reorganization of the motor cortex. It is not clear if the physiological change induced by BoNT therapy had any correlation with the clinical improvement. In addition, it is not clear if the change in motor cortex excitability ultimately affects the corticospinal drive to the dystonic muscles.

In this study, the investigators will focus on the physiological effects of BoNT using broader TMS measures of motor cortex excitability. The central hypothesis is that BoNT modulates the motor cortex excitability and the corticospinal drive to the muscles and that these physiological effects of BoNT will have a clear correlation with the clinical response. To test this hypothesis, the investigators plan to measure the corticospinal drive to dystonic muscles using electromyographic (EMG) spectral analysis. They will record the clinical outcome with the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) which is a standardized validated rating scale for PCD.

The first and second aim will focus on the physiological aspects of BoNT therapy in PCD. The investigators plan to determine the cortical and corticospinal physiologic changes at the time of peak BoNT effects (BoNT ON) which are typically seen around 4-8 weeks after the injections and at the time of wearing off related to BoNT therapy which will correspond to the time of the next injection cycle (BoNT OFF). The third aim will help the investigators understand the physiological differences between clinical responders and non-responders. Healthy controls will be enrolled for normative physiological data. The main significance of this study is advancement of physiological knowledge related to BoNT therapy in subjects with PCD.

Aim 1:

To determine the effect of BoNT therapy on the motor cortex excitability in PCD.

TMS measures (such as SICI, ICF,...) will be collected using standardized protocols at the time of peak BoNT effects (BoNT ON) and at the time of trough BoNT effects (BoNT OFF).

Hypothesis 1:

The TMS measures will be normalized to healthy controls at the time of peak BoNT effects and these effects will reverse once the BoNT effects wear off.

Aim 2:

To determine the effects of BoNT therapy on the corticospinal drive to the PCD muscles.

EMG spectral analysis for the auto-spectral peak of 4-7 Hertz (Hz) at the sternocleidomastoid (SCM) and the 10-12 Hz coherence between the SCM and the splenius capitis (SPL) will be used at the time of peak (BoNT ON) and trough BoNT effects (BoNT OFF).

Hypothesis 2:

The coherence between SPL and SCM muscles will be lost at the time of peak BoNT effects. There will be a re-appearance of the auto-spectral peak in SPL muscle as seen in healthy controls. These spectral analysis changes will reverse as the BoNT effects wear off during trough.

Aim 3:

To determine the correlation between the physiological measures (TMS and EMG measures) during peak BoNT effects and the clinical scores.

Hypothesis 3:

The change in TMS measures and EMG spectral findings at the time of peak BoNT effects will correlate with the change in clinical score on the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale.

ELIGIBILITY:
Subject inclusion criteria:

* Diagnosis: PCD
* Receiving BoNT at the University of Florida (UF)

Subject exclusion criteria:

* Secondary torticollis
* Pregnancy
* Active seizure disorder
* Presence of metallic body such as pacemaker, implants, metal rods and hearing aid

Control inclusion criteria:

* Age 21-80 years

Control exclusion criteria:

* Any form of torticollis
* Pregnancy
* Active seizure disorder
* Presence of metallic body such as pacemaker, implants, metal rods and hearing aid

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Changes in TMS measures | Baseline, BoNT ON (around 6 weeks), BoNT OFF (around 12 weeks) for Arm 1; Arm 2 measured only at baseline
Changes in EMG measures | baseline, BoNT ON (around 6 weeks), BoNT OFF (around 12 weeks) for Arm 1; Arm 2 measured only at baseline

SECONDARY OUTCOMES:
Changes in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | 0, BoNT ON (around 6 weeks), BoNT OFF (around 12 weeks) for Arm 1 only
  Clinical measurement of cervical dystonia

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes